CLINICAL TRIAL: NCT00900237
Title: A Phase I, Single Centre, Open, Randomised, Parallel Study to Evaluate the Pharmacokinetics and Tolerability of Multiple Doses of Eslicarbazepine Acetate and Oxcarbazepine in Healthy Subject
Brief Title: Study to Evaluate Pharmacokinetics and Tolerability of Multiple Doses of Eslicarbazepine Acetate and Oxcarbazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-127
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Partial Epilepsy
Keywords: Partial; Epilepsy; Eslicarbazepine acetate; Pharmacokinetics; Tolerability
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — eslicarbazepine acetate; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eslicarbazepine acetate (Active Comparator): Eslicarbazepine acetate (ESL) 600 mg QD morning from Day 1-3 and 1200 mg ESL QD morning from Day 4-9
  Interventions: Drug: Eslicarbazepine acetate
- Oxcarbazepine (Active Comparator): Oxcarbazepine 300 mg BID from Day 1-3 and oxcarbazepine 600mg BID from Day 4-9
  Interventions: Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Eslicarbazepine acetate — Oral administration 600 mg QD morning from Day 1-3 and 1200 mg from Day 4-9
  Other Names: BIA 2-093
  Arms: Eslicarbazepine acetate
Drug: Oxcarbazepine — Oxcarbazepine 300 mg BID from Day 1-3 (morning and evening) and oxcarbazepine 600mg BID from Day 4-9 (morning and evening, only morning dose on Day 9)
  Other Names: Trileptal; Trexapin; 10,11-Dihydro-10-oxo-5 H -dibenz(b,f)azepine-5-carboxamide
  Arms: Oxcarbazepine

SUMMARY:
This purpose of this study is to measure the concentrations of two anti-epileptic drugs (Eslicarbazepine acetate and oxcarbazepine) and their metabolites in the cerebrospinal fluid and blood plasma of healthy subjects and also to assess how these drugs are tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Aged 18-55 years
* Body mass index (18.5-29 kg/m3)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luc Cavens, MD, Principal Investigator — SGS LSS Clinical Pharmacology Unit Antwerpen
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerpen, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eslicarbazepine Acetate | Oxcarbazepine
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eslicarbazepine Acetate | Oxcarbazepine | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Plasma Concentration in Plasma and Cerebral Spinal Fluid
Description: Cmax - Maximum plasma concentration CSF - Cerebral Spinal Fluid Oxcarbazepine, BIA 2-194 and BIA 2-195 are active metabolites of Eslicarbazepine Acetate.
Time Frame: Day 9 - Pre-dose; 0.5h; 1h; 1.5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h; 24h
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eslicarbazepine Acetate | Oxcarbazepine
Number analyzed (Participants) | 7 | 7
ng/mL
  Cmax (BIA 2-194) plasma | 23932 (6630) | 16162 (2662)
  Cmax (BIA 2-195) plasma | 886 (235) | 4039 (613)
  Cmax (Oxcarbazepine) plasma | 245 (72.6) | 1990 (941)
  Cmax (BIA 2-194) CSF | 7559 (1050) | 7566 (912)
  Cmax (BIA 2-195) CSF | 538 (145) | 2146 (327)
  Cmax (Oxcarbazepine) CSF | 93.2 (27.0) | 448 (109)

2. Primary Outcome: AUC0-t AUC From Time Zero to the Last Sampling Time
Description: AUC0-t - area under the concentration versus time curve (AUC) from time zero to the last sampling time at which concentrations were at or above the limit of quantification CSF - cerebrospinal fluid Oxcarbazepine, BIA 2-194 and BIA 2-195 are active metabolites of Eslicarbazepine Acetate.
Time Frame: Day 9 - Pre-dose; 0.5h; 1h; 1.5h; 2h; 3h; 4h; 6h; 8h; 12h; 16h; 24h
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Eslicarbazepine Acetate | Oxcarbazepine
Number analyzed (Participants) | 7 | 7
ng.h/mL
  AUC0-t (BIA 2-194) plasma | 340123 (70412) | 164726 (29904)
  AUC0-t (BIA 2-195) plasma | 18743 (4620) | 39034 (7094)
  AUC0-t (Oxcarbazepine) plasma | 3377 (762) | 7135 (2561)
  AUC0-t (BIA 2-194) CSF | 154509 (22495) | 86187 (9545)
  AUC0-t (BIA 2-195) CSF | 11791 (2909) | 23996 (3495)
  AUC0-t (Oxcarbazepine) CSF | 1522 (287) | 2485 (400)

ADVERSE EVENTS:
Arm/Group | Eslicarbazepine Acetate | Oxcarbazepine
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eslicarbazepine Acetate (N=7) | Oxcarbazepine (N=7)
Dizziness (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 2 | 7
Somnolence (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 2 | 1
Memory impairment (Nervous system disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 5
Stomach discomfort (Gastrointestinal disorders) | 0 | 3
Hypoesthesia oral (Gastrointestinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Fatigue (General disorders) | 2 | 5
Vision blurred (Eye disorders) | 0 | 3
Nasopharyngitis (Infections and infestations) | 0 | 2
Postlumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other